CLINICAL TRIAL: NCT04236401
Title: Cold Knife Versus Monopolar Electrosurgery for Abdominal Incisions ( Clinical Trial )
Brief Title: Cold Knife Versus Monopolar Electrosurgery in Abdominal Incisions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Shimaa Esmail Borhamy Khalaf, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Electrosurgery
Record Dates: First submitted 2019-12-23; First posted 2020-01-22 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Electrosurgery Versus Scalpel
Keywords: electrosurgery; scalpel; abdominal incision
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electrosurgery will be used inanterior abdominal wall incision (Other): to perform benign gynecological conditions , surgeon will need to open anterior wall electrosurgically.
  Interventions: Procedure: electrosurgery will be used for abdominal incision
- scalpel will be used in abdominal wall incision (Other): to perform benign gynecological conditions , surgeon will need to open anterior wall sharply.
  Interventions: Procedure: scalpel will be used for abdominal incision

INTERVENTIONS:
Procedure: electrosurgery will be used for abdominal incision — electrosurgery will be used to open anterior abdominal wall and electrosurgery will be used for heamostasis also
  Arms: electrosurgery will be used inanterior abdominal wall incision
Procedure: scalpel will be used for abdominal incision — scalpel will be used for abdominal wall incision and thread will be used for haemostsis
  Arms: scalpel will be used in abdominal wall incision

SUMMARY:
the aim of work is to compare the early postoperative and late term wound complication rates between the scalpel and electrosurgery in patients with benign gynecological conditions undergoing abdominal incisions.

DETAILED DESCRIPTION:
• Study Hypothesis: - Using electrosurgery decrease incision blood loss, decrease postoperative pain, decrease wound time incision, decrease analgesia requirements, doesn't increase wound sepsis.

Type of study: - Randomized controlled trial study (parallel group study with 1:1 randomization) will be conducted at gynecology department of Alzhraa University Hospital of faculty of Medicine for girls - Cairo within 1 year according to sample size. A computer randomization will be generated and held with one of the experimenter, and (n) of black and red card will be used for allocation concealment.

Participants at morning of the operation will be given information about the study aims and written consent will be taken.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective gynecological abdominal surgeries for benign diseases
* willing to participate in the study.
* The participants will receive 2 gm cephalosporines preoperative per hospital policy.

Exclusion Criteria:

* History of receiving antibiotics during the preceding 7 days,
* chronic medical illness like diabetes, asthma or tuberculosis,
* patients have anemia,
* surgically scarred tissues,
* Immuno-compromised patients,
* pregnant patients,
* patients with pacemaker device,
* patients on anticoagulants therapy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Wound incision time | at the beginning of each surgery
  measure time needed to open anterior abdominal wall in minutes by stopwatch
Wound infection | after surgery till primary healing of the wound, an average of 15 days after operation
  rate of infection in wound after surgery as inflammation, seroma, heamatoma, gapping, sepsis or fever

SECONDARY OUTCOMES:
Postoperative pain (pain score 2-4 hr postoperative). | during first 4 hours after surgery
  using Visual Analogue Scale; the higher scores mean worse outcome
Amount of Analgesia needed during 1st 12 hr after surgery . | first 12 hours after surgery
  dose of analgesia needed
Wound-related blood loss | after opening anterior abdominal wall during each surgery
  by weighing towel before and after abdominal wall incision / grams
number of participants with bad scar formation or keloid | through study completion, an average of 1.25 year
  scar condition evaluation after complete healing of the wound. early healing after 15 days of the surgery and after complete healing after 45 days of the surgery